CLINICAL TRIAL: NCT02296346
Title: A Randomized, Controlled, Open-Label Study to Evaluate the Efficacy of Extracorporeal Photopheresis (ECP) Versus Corticosteroids in the Treatment of Patients With Secondary Progressive Multiple Sclerosis (SPMS)
Brief Title: Open-Label Study to Evaluate the Efficacy of ECP in Secondary Progressive Multiple Sclerosis
Acronym: MSECP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment/PI relocated. New site couldn't reach agreement with manufacturer
Sponsor: University of Utah (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Daniel Couriel, M.D., University of Utah
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00083301
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Methylprednisolone Hemisuccinate; Adrenal Cortex Hormones; Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroid arm (Active Comparator): Patients will receive 1 gram of IV SoluMedrol over 1 hour, once every month for 12 months.
  Interventions: Drug: SoluMedrol
- Extracorporeal Photopheresis (Experimental): Patient will receive an Extracorporeal Photopheresis treatment at a set frequency over the course of 1 year. The treatment takes about 2-3 hours per session to complete. The treatment schedule is as follows:
  ECP will be administered according to the following schedule:
  Study Arm: Weeks 1-8: 3 times per week Weeks 9-16: Twice per week Weeks 17-36: Treatment on two consecutive days every 2 weeks (or optionally, one treatment per week) Weeks 37-43: Once every 2 weeks Weeks 44-52: Once every 4 Weeks
  Interventions: Device: Extracorporeal Photopheresis

INTERVENTIONS:
Drug: SoluMedrol — Infusion of drug subcutaneously, once a month.
  Other Names: Corticosteroids
  Arms: Corticosteroid arm
Device: Extracorporeal Photopheresis — This intervention is the placement of up to two IV's to extract your blood as a set volume, separate out the white cells and return the red cells to your body. Then the white cells are treated with a drug called UVADEX (methoxsalen), excited by a UV light and returned to your body. Once IV is to withdraw your blood and the other is to return your blood to your body.
  Other Names: ECP; Cellex machine; Therakos
  Arms: Extracorporeal Photopheresis

SUMMARY:
In this research study, the investigators will determine whether a procedure called Extracorporeal Photopheresis (ECP) is helpful in preventing progression of disability in people with SPMS when compared to monthly corticosteroid infusions. This study will determine whether ECP has an effect on inflammatory cells in people with SPMS and whether it has a beneficial therapeutic effect.

DETAILED DESCRIPTION:
This is a Phase II randomized, open-label study to evaluate the efficacy of extracorporeal photopheresis (ECP) versus IVMP on disability progression in subjects with SPMS. At the initial screening visit, an extensive medical history will be obtained and a detailed neurological examination will be performed to determine eligibility. Subjects who meet eligibility criteria will be enrolled in one of two study arms. Subjects will be randomized at a 1:1 ratio to receive ECP (study arm) or active treatment with intravenous methylprednisolone pulses (control arm) administered every 4 Weeks (1 gram per infusion) for 52 weeks.

ECP will be administered according to the following schedule:

Study Arm: Weeks 1-8: 3 times per week Weeks 9-16: Twice per week Weeks 17-36: Treatment on two consecutive days every 2 weeks (or optionally, one treatment per week) Weeks 37-43: Once every 2 weeks Weeks 44-52: Once every 4 Weeks

All subjects, including patients who receive corticosteroids, will be evaluated using the MSFC tool at baseline and every 3 months through 2 years. They will also be scored using the EDSS at baseline and every 3 months through 2 years. Subjects in the control arm will be evaluated by MSFC and EDSS during the week prior to their next intravenous methylprednisolone infusion and every three months from baseline through two year mark. Blood will be collected for immune function (cytokines) testing at baseline, and months 3, 6, 9 and 12. MRI will be done at baseline as well as months 6 and 12 following initiation of treatment; if the disability measurements are stable or improved at any point in time, then ECP will be continued per protocol..

Patients in the ECP arm should have all of their treatments with the CELLEX ® System. Patients randomized to the ECP arm must receive their treatment within 5 days of baseline visit.

In the ECP process, UVADEX ® (methoxsalen) Sterile Solution will be injected directly the recirculation bag of the extracorporeal circuit after completion of the buffy coat collection. The dose of UVADEX® (methoxsalen) Sterile Solution will be calculated based on the standard treatment volume formula.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SPMS based on the Recommended Diagnostic Criteria for MS and clinical course.
* Demonstrate EDSS scores between 3 to 6.5 at screening.
* Documented EDSS progression in the 2 years prior to screening of 1 point or greater for patients with an EDSS score less than 6 at baseline, and greater than or equal to 0.5
* Documented absence of clinical relapse within 2 years of screening
* Age ≥ 18 ≤ 75 years
* Weight > 40≤ 150 kg.
* Absolute Neutrophil count ≥ 2,000 per μL
* Hematocrit ≥ 28 % and platelet count > 100,000 per μL (with or without transfusion support)
* Willingness to use at least 1 reliable method of birth control (e.g. abstinence, oral contraceptives, intrauterine devices, barrier method with spermicide, or surgical sterilization) throughout the study for all men and women of childbearing potential
* Willingness to participate in all study visits and procedures, as outlined in the informed consent
* Patients able to give informed consent.
* Patients must have adequate peripheral venous access to initiate ECP therapy.

Exclusion Criteria:

* Absolute medical contraindication to corticosteroid treatment
* Absolute medical contraindication to receive ECP
* Clinical relapse within 2 years of screening
* Laboratory evidence of any of the following:

  * WBC < 2,000 cells per uL
  * Serum transaminase levels > x 2 UNL
  * HgbA1C > 6%
* Concurrent diagnosis of a neurological condition or autoimmune disease other than MS
* Evidence of known infection with human immunodeficiency virus (HIV) or active (not including latent) Hepatitis B (laboratory testing is not required if virus status is already known)
* Uncontrolled infection requiring treatment at study entry
* Hypersensitivity or allergy to psoralen (methoxsalen)
* Hypersensitivity or allergy to both heparin and citrate products (If hypersensitive or allergic to only one of these products, exclusion does not apply)
* Inability to tolerate fluid changes associated with ECP (e.g. inadequate renal, hepatic, pulmonary and cardiac function leading to enable patient to tolerate extracorporeal volume shifts associated with ECP)
* Presence of aphakia or photosensitive disease (systemic lupus erythematosis, porphyrias, albinism, etc.)
* Women who are pregnant and/or lactating.
* Use of any investigational drug/treatment at the time of enrollment or within the previous 60 days, or five elimination half-lives, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
* Initiation of dalfampridine or change in the dose of dalfampridine within 6 months prior to randomization
* Treatment with any of the medications or procedures listed below:

  * Glatiramer acetate, interferon-beta, fingolimod, teriflunomide or dimethylfumarate within 3 months prior to randomization
  * Natalizumab within 6 months prior to randomization
  * Cyclophosphamide within 1year prior to randomization
  * Mitoxantrone within 2 years prior to randomization
  * Rituximab, ofatumumab, ocrelizumab, cladribine, daclizumab within 2 years prior
  * Intravenous immunoglobulin within 6 months prior to randomization
  * Plasmapheresis within 1 year prior to randomization
  * Corticosteroids within 3 months prior to screening
* Inability to undergo MRI scans
* Contraindication to gadolinium due to past allergic, hypersensitive or adverse reaction or impaired renal function
* Any other disease or condition which, in the opinion of the investigator, could interfere with participation in the study according to the study protocol, or with the ability of the patients to cooperate and comply with study procedures.
* Poor venous access
* Previous history of skin cancer, leukemia/lymphoma/myeloma or bone marrow transplant.
* History of cataracts
* Patients taking Coumadin who are unable to switch from oral anticoagulants to enoxaparin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2018-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Segal, MD, Principal Investigator — University of Michigan, Director of Multiple Sclerosis Center; Daniel Couriel, MD, Principal Investigator — University of Utah, Huntsman Cancer Institute, Internal Medicine
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Corticosteriod Arm: Patients will receive 1 gram of IV SoluMedrol over 1 hour, once every month for 12 months.
  SoluMedrol: Infusion of drug subcutaneously, once a month.
- Extracorporeal Photopheresis: Patient will receive an Extracorporeal Photopheresis treatment at a set frequency over the course of 1 year. The treatment takes about 2-3 hours per session to complete. The treatment schedule is as follows:
  ECP will be administered according to the following schedule:
  Study Arm: Weeks 1-8: 3 times per week Weeks 9-16: Twice per week Weeks 17-36: Treatment on two consecutive days every 2 weeks (or optionally, one treatment per week) Weeks 37-43: Once every 2 weeks Weeks 44-52: Once every 4 Weeks
  Extracorporeal Photopheresis: This intervention is the placement of up to two IV's to extract your blood as a set volume, separate out the white cells and return the red cells to your body. Then the white cells are treated with a drug called UVADEX (methoxsalen), excited by a UV light and returned to your body. Once IV is to withdraw your blood and the other is to return your blood to your body.
Period: Overall Study
Arm/Group | Corticosteriod Arm | Extracorporeal Photopheresis
Started | 7 | 6
Completed | 2 | 0
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corticosteriod Arm | Extracorporeal Photopheresis | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Multiple Sclerosis Functional Composite (MSFC) [Mean (Full Range); unit: MSFC z-score] — MSFC score is a composite score calculated from 3 tests: 1) Timed 25-Foot walk (leg function); 2) 9-Hole Peg Test (arm function); and 3) Paced Auditory Serial Addition Test (cognitive function). The results are combined to create a single score (the MSFC Z-Score) to measure performance and change over time in subjects with MS. MSFC Z-score = {Z arm + Z leg + Z cognitive} / 3.0. A positive score indicates that, on average, an individual performed better than the reference population and a negative score indicates that, on average, an individual performed worse than the reference population.
  MSFC z-score | 0.2410 [-0.361 to 0.6419] | -0.2335 [-0.842 to 0.7335] | 0.0022 [-0.842 to 0.7335]
Expanded Disability Status Scale (EDSS) [Mean (Full Range); unit: EDSS Score] — The Expanded Disability Status Scale (EDSS) is used to quantify disability due to symptoms of MS and to track changes in disability status over time. Scores range from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). Scores are determined by performing a neurological exam and given in increments of 0.5.
  EDSS Score | 6 [4.5 to 6.5] | 5.92 [4.0 to 6.5] | 5.96 [4.0 to 6.5]

OUTCOME MEASURES:

1. Primary Outcome: Multiple Sclerosis Functional Composite (MSFC) Z-score and Expanded Disability Status Scale (EDSS)
Description: MSFC score is a composite score calculated from 3 tests: 1) Timed 25-Foot walk (leg function); 2) 9-Hole Peg Test (arm function); and 3) Paced Auditory Serial Addition Test (cognitive function). The results are combined to create a single score (the MSFC Z-Score) to measure performance and change over time in subjects with MS. MSFC Z-score = {Z arm + Z leg + Z cognitive} / 3.0. A positive score indicates that, on average, an individual performed better than the reference population and a negative score indicates that, on average, an individual performed worse than the reference population.
  The Expanded Disability Status Scale (EDSS) is used to quantify disability due to symptoms of MS and to track changes in disability status over time. Scores range from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). Scores are determined by performing a neurological exam and given in increments of 0.5.
Time Frame: 1 year
Population: Baseline MSFC and EDSS scores were captured for all 13 subjects, however some subjects withdrew immediately after baseline. Withdrawal of additional subjects continued from that point. Only 1 patient from the ECP arm made it to the 12 month visit. Four patients from the CS arm made it to 12 mos, however 1 of the 4 declined the MSFC tests.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- ECP Arm: Study participants assigned to ECP treatment
- Corticosteroid Arm: Study participants assigned to corticosteroid treatment
Arm/Group | ECP Arm | Corticosteroid Arm
Number analyzed (Participants) | 1 | 4
score on a scale
  EDSS Score | 6 [6 to 6] | 6.25 [6 to 6.5]
  MSFC Z-Score: number analyzed (Participants) | 1 | 3
  MSFC Z-Score | 1.1031 [1.1031 to 1.1031] | 0.6751 [0.4914 to 0.9504]

2. Secondary Outcome: Immunological Parameters in Relation to SPMS
Description: Changes in immunological parameters that occur following initiation of ECP or corticosteroids and any relevant correlation with clinical outcomes
Time Frame: 2 year
Population: Due to low enrollment numbers and a high dropout rate, there was insufficient data to analyze and correlate treatment with clinical outcomes. Only 2 subjects continued to the 24 month completion, both were corticosteroid patients. No ECP subjects made it to 24 mos. Therefore, there was no analysis performed on the 2 year data.
Arm/Group | Corticosteriod Arm | Extracorporeal Photopheresis
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on study participants from baseline visit to study completion, approximately 2 years.
Arm/Group | Corticosteriod Arm | Extracorporeal Photopheresis
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/6
Other Adverse Events (participants affected / at risk) | 6/7 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteriod Arm (N=7) | Extracorporeal Photopheresis (N=6)
Suicide (Psychiatric disorders) | 0 (0) | 1 (1) — Subject committed suicide shortly after withdrawing from the trial and experiencing disease progression/worsening of MS symptoms.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corticosteriod Arm (N=7) | Extracorporeal Photopheresis (N=6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5) — Subject experienced pneumonia on 4 separate occasions; Ruled expected and unlikely to be attributed to trial.
Poor Venous Access (Vascular disorders) | 0 (0) | 1 (1) — Ruled Unexpected and Related.
Nocturnal Hypoxia (on PSG) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Ruled unexpected and unlikely to be related.
Iron Deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Ruled expected and probably related.
Low Hematocrit Requiring Transfusion of 1 unit PRBC (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Ruled unexpected and probably related.
Acute blood loss not requiring transfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Ruled unexpected and probably related.
Catheter Line Crack (Vascular disorders) | 0 (0) | 1 (1) — Ruled unexpected and related.
"Jittery" Sensation during treatment (General disorders) | 1 (1) | 0 (0) — Subject reported sensation during infusion treatment; Ruled expected and related.
Dizziness (General disorders) | 0 (0) | 1 (1) — Ruled expected and probably related to treatment.
Urinary tract infection (Renal and urinary disorders) | 3 (5) | 0 (0) — Multiple subjects experienced urinary tract infections throughout the trial. All ruled expected and unlikely to be related.
Acute Cystitis without Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) — Ruled unexpected and unlikely to be related.
Mild Hives (General disorders) | 0 (0) | 1 (1) — Subject experienced mild hives during an MRI; Ruled unexpected and probably related.
Knee Pain and Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Ruled unexpected and unlikely to be related.
Chest pain (General disorders) | 1 (1) | 0 (0) — Ruled unexpected and unlikely to be related to trial.
Obstructive Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — Ruled unexpected and unlikely to be related in both subjects.
Mild Concussion (Nervous system disorders) | 1 (1) | 0 (0) — Ruled unexpected and unlikely to be related to trial.
Low Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Ruled expected and probably related to trial.
Petechial Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject experienced petechial rash on left chin; Ruled unexpected and unlikely to be related.
Infiltrated IV with treatment (Vascular disorders) | 1 (1) | 0 (0) — AE ruled expected and probably related.
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — In both subjects, infections were ruled expected and unlikely to be related.
Spinal Vertebral Lesions (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject noted to have 3 new spinal vertebral lesions on MRI. AE ruled expected and unlikely to be related.
Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject experienced swelling in left calf. AE ruled unexpected and unlikely to be related.
Anxiety Attacks (Psychiatric disorders) | 0 (0) | 1 (1) — Subject experienced intermittent anxiety attacks; Ruled unexpected and unlikely to be related to trial.
Groin Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) — AE ruled unexpected and unlikely to be related.
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) — AE ruled expected and unlikely to be related.
Pressure Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Stage 1 Pressure Ulcer in right foot. Ruled unexpected and unlikely to be related to trial
Ear Congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Ruled unexpected and unlikely to be related to trial
Infusion Reaction (General disorders) | 1 (1) | 0 (0) — Subject experienced reaction while receiving infusion of Rituximab. AE ruled expected and unlikely to be related to trial.

LIMITATIONS AND CAVEATS:
Analysis of the data in this study was severely limited by the high dropout rate and low enrollment numbers. Given that only 2/13 participants completed the study, we do not have enough outcome data to complete a meaningful analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT02296346/Prot_SAP_000.pdf